CLINICAL TRIAL: NCT02215707
Title: A Clinical Trial of the PfSPZ Vaccine Administered by Direct Venous Inoculation in Healthy Malaria-Naïve Adults: Heterologous vs. Homologous Controlled Human Malaria Infection and Reduction in Number of Doses
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanaria Inc. (Industry)
Collaborators: Naval Medical Research Center (U.S. Federal Agency); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); Military Infectious Diseases Research Program (MIDRP) (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WRAIR #2080; NMRC.2014.004 (Other: Naval Medical Research Center); WRAIR #2080 (Other: Walter Reed Army Institute of Research)
Record Dates: First submitted 2014-08-01; First posted 2014-08-13 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2015-11

CONDITIONS: Malaria
Keywords: PfSPZ Vaccine; Plasmodium falciparum; Malaria; Controlled Human Malaria Infection (CHMI)
MeSH Terms: conditions — Malaria; Malaria, Falciparum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Group 1 (Experimental): Group 1: 5 doses of 2.7x10^5 PfSPZ Vaccine; homologous 3D7 CHMI
  Grp 1 (n=15) gets 5 doses of 270,000 PfSPZ per dose (4 doses at 4 wk intervals, 2 month delay before 5th dose) by DVI. Grps 1 and 2 start immunizations together.
  1 subj in each of Grps 1 and 2 will be immunized approx 24 hrs before rest of grp ("pilot subjects"). For Grp1/Grp 2 pilot subjects: 1st subject will be immunized, observed on site for minimum 1 hr; the 2nd subject may be immunized, will also be observed for minimum 1 hr. If no safety concerns are identified after 24 hrs that trigger the stopping rules, then rest of subjects in Grps 1 and 2 will be immunized.
  Approx 3 wks after final dose, Grps 1 and 3 will undergo homologous CHMI (Pf3D7 strain) with 6 Infectivity Controls. Approx 24 wks after last dose, Grps 1 and 3 will undergo 2nd homologous CHMI (3D7) with 6 Infectivity Controls. Subjects will be followed for 8 wks after last CHMI for safety purposes.
  Interventions: Biological: PfSPZ Vaccine
- Group 2 (Experimental): Grp 2: 5 doses of 2.7x10^5 PfSPZ Vaccine; heterologous 7G8 CHMI
  Grp 2 (n=15) gets 5 doses of 270,000 PfSPZ/dose (4 doses at 4wk intervals, 2 month delay before 5th dose) by DVI. Grps 1 / 2 start immunizations together.
  1 subj in each of Grps 1 / 2 will be immunized approx 24 hrs before rest of grp ("pilot subjects"). For Grp1/ 2 pilot subj: 1st subj will be immunized, observed on site for min 1 hr; 2nd subj may be immunized, will also be observed for min 1 hr. If no safety concerns after 24 hrs that trigger stopping rules, then rest of Grps 1 / 2 will be immunized.
  Approx 3 wks after final dose, Grps 1/3 have homologous CHMI; 2-3 days later, Grp 2 will undergo heterologous CHMI (Pf7G8) with 6 Infectivity Controls. Approx 24 wks after last dose, Grps 1/3 have 2nd homologous CHMI; 2-3 days later, Grp 2 will undergo 2nd heterologous CHMI (7G8 strain) with 6 Infectivity Controls. Subj will be followed for 8 wks after last CHMI for safety purposes.
  Interventions: Biological: PfSPZ Vaccine
- Group 3 (Experimental): Grp 3 (n=15) will receive 3 doses by DVI of 450,000 PfSPZ/dose (of PfSPZ Vaccine) at 8 wk intervals (starting approx. 4 wks after Grps 1 and 2 get 1st immunization).
  3 subjects in Grp 3 will be immunized approx 24 hrs prior to rest of grp ("pilot subjects"). The 3 subjects will be immunized sequentially with min 2 hr observation period between subjects (and a 2 hr observation of 3rd subject as well). If no safety concerns identified in pilot subjects after 24 hours that trigger the stopping rules, the rest of subjects in Grp 3 will be immunized as scheduled.
  Approx 3 wks after final dose, Grps 1 and 3 will undergo homologous CHMI (3D7 strain) with 6 Infectivity Controls. Approx 24 wks after last dose, Grps 1 and 3 will undergo 2nd homologous CHMI (3D7) with 6 Infectivity Controls. Subjects will be followed for 8 wks after last CHMI for safety purposes.
  Interventions: Biological: PfSPZ Vaccine
- CHMI Controls.1 (No Intervention): n = 6, infectivity controls for 1st homologous CHMI (3D7) occurring approximately 3 weeks after final immunization of Groups 1 and 3. This group does not receive the PfSPZ Vaccine.
- CHMI Controls.2 (No Intervention): n = 6, infectivity controls for 1st heterologous CHMI (7G8) occurring approximately 3 weeks after final immunization of Group 2. This group does not receive the PfSPZ Vaccine.
- CHMI Controls.3 (No Intervention): n = 6, infectivity controls for 2nd homologous CHMI (3D7) occurring approximately 24 weeks after final immunization of Groups 1 and 3. This group does not receive the PfSPZ Vaccine.
- CHMI Controls.4 (No Intervention): n = 6, infectivity controls for 2nd heterologous CHMI (7G8) occurring approximately 24 weeks after final immunization of Group 2. This group does not receive the PfSPZ Vaccine.

INTERVENTIONS:
Biological: PfSPZ Vaccine — Suspension of metabolically active, non-replicating (live), radiation-attenuated, purified, cryopreserved, aseptic Plasmodium falciparum (Pf) sporozoites (SPZ)
  Arms: Group 1; Group 2; Group 3

SUMMARY:
This is an open-label evaluation of the safety, tolerability immunogenicity and efficacy of the PfSPZ Vaccine administered by Direct Venous Inoculation (DVI) in healthy, malaria-naïve subjects. There will be 3 groups and a total of 69 subjects (45 immunized subjects and 24 infectivity controls).

DETAILED DESCRIPTION:
Group 1 (n=15) and Group 2 (n = 15) subjects will receive five doses by DVI of 2.7 x 10^5 PfSPZ per dose (4 doses at 4 week intervals and the 5th dose 8 weeks after the fourth dose). Group 3 (n = 15) will receive 3 doses by DVI of 4. 5 x 10^5 PfSPZ/dose at 8 week intervals. Subjects who complete all immunizations will receive a total 13.5 x 10^5 PfSPZ. Protective efficacy will be assessed by Controlled Human Malaria Infection (CHMI) by exposure to the bites of five Pf-infected mosquitoes. Groups 1 and 3 (n = 30) will undergo each of two CHMIs at the same time with mosquitoes infected with PfSPZ (3D7) (homologous) along with 6 Infectivity Controls. Group 2 will undergo each of two CHMIs separately with mosquitoes infected with PfSPZ (7G8) (heterologous) along with 6 Infectivity Controls. CHMI will occur at approximately 2 to 3 weeks and 24 weeks after the final immunization. Subjects may proceed to CHMI provided they have received no fewer than three scheduled immunizations. Immunized subjects may participate in the second CHMI whether or not they were protected in the first CHMI; boosting of immune responses in CHMI #1 may lead to protection in CHMI #2.

One subject in each of Groups 1 and 2 and 3 subjects in Group 3 will be immunized approximately 24 hours prior to the rest of the group (referred to as "pilot subjects"). For the Group1/Group 2 pilot subjects: the first subject will be immunized and observed on site for a minimum of one hour; at this point, the second subject may be immunized and he/she will also be observed for a minimum of one hour. For Group 3: the three subjects will be immunized sequentially with a minimum 2 hour observation period between subjects (and a two hour observation of the third subject as well). If there are no safety concerns identified in the pilot subjects after 24 hours that trigger the stopping rules, then the rest of subjects in Groups 1, 2 and 3 will be immunized as scheduled. Subjects in Group 3 will receive their first immunization approximately 4 weeks after subjects in Groups 1 and 2 receive their first immunizations. Subjects will be followed for 8 weeks after the last CHMI for safety purposes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults (male or non-pregnant female) 18 - 45 years of age, inclusive.
* Able and willing to participate for the duration of the study.
* Able and willing to provide written (not proxy) informed consent.
* Women of childbearing potential must agree to use effective means of birth control (e.g. oral or implanted contraceptives, IUD, female condom, diaphragm with spermicide, cervical cap, abstinence, use of a condom by the sexual partner or sterile sexual partner) during the entire study. Women with a history of surgical or chemical sterilization (e.g. tubal ligation, hysterectomy, other) must provide written documentation of infertility from a Primary Care Provider.
* Willing to refrain from blood donation (except as required in this study) for 3 years following CHMI.
* Agree not to travel to a malaria endemic region during the entire course of the trial.

Exclusion Criteria:

* Any history of malaria infection, or travel to a malaria endemic region within 6 months prior to first immunization.
* History of long-term residence (>5 years) in area known to have significant transmission of P. falciparum.
* Has evidence of increased cardiovascular disease risk (defined as > 10%, 5 year risk) as determined by the method of Gaziano [Gaziano, 2008]. Risk factors include sex, age, systolic blood pressure (mm Hg), smoking status, body mass index (BMI, kg/mm2), and reported diabetes status.
* Positive HIV, HBsAg or HCV serology.
* Positive sickle cell screening test.
* An abnormal electrocardiogram, defined as one showing pathologic Q waves and significant ST-T wave changes; left ventricular hypertrophy; any non-sinus rhythm including isolated premature ventricular contractions, but excluding isolated premature atrial contractions; right or left bundle branch block; or advanced (secondary or tertiary) A-V heart block.
* Current use of systemic immunosuppressant pharmacotherapy.
* Current significant medical condition (cardiovascular, hepatic, renal, or hematological) or evidence of any other serious underlying medical condition identified by medical history, physical examination, or laboratory examination.
* History of a splenectomy.
* History of neurologic disorder (including seizures) or migraine headache.
* History of psychiatric disorders (such as personality disorders, anxiety disorders, or schizophrenia) or behavioral tendencies (including active alcohol or drug abuse) discovered during the screening process that in the opinion of the investigator would make compliance with the protocol difficult.
* Plan for surgery between enrollment and CHMI.
* Females who are pregnant or nursing, females who plan on becoming pregnant or plan to nurse during the study period.
* Known allergy to any component of the vaccine formulation, history of anaphylactic response to mosquito-bites, or any history of anaphylactic reaction, retinal or visual field changes, or known allergy to anti-malarials including chloroquine phosphate, atovaquone/proguanil (Malarone®), or artemether/lumefantrine (Coartem®)
* Receipt of another investigational vaccine or drug within 30 days prior to the first immunization, or plan to participate in another investigational vaccine/drug research during or within 1 month following participation in this study.
* Receipt of more than three other vaccines within 60 days prior to the screening visit, or plan to receive more than three other vaccines during or within 1 month following participation in this study.
* Personal beliefs that prohibit the receiving of vaccine product containing human serum albumin within the diluent (vaccine recipients only).
* Use or planned use of any drug with anti-malarial activity that would coincide with the periods of immunization or CHMI.
* History of psoriasis or porphyria, which may be exacerbated after treatment with chloroquine.
* Anticipated use of medications known to cause drug reactions with chloroquine, atovaquone-proguanil (Malarone®), or artemether/lumefantrine (Coartem®) such as cimetidine, metoclopramide, antacids, and kaolin.
* History of any other illness or condition which, in the investigator's judgment, may substantially increase the risk associated with the subject's participation in the protocol or compromise the scientific objectives.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2014-06; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Incidence and type of adverse events (including breakthrough infections), vital signs, clinical laboratory assessments, physical examination findings. | Day of immunization through week 52
Evidence of vaccine-mediated protection against CHMI 2-3 weeks and 24 weeks after last immunization in Groups 1, 2, and 3, preventing blood stage infection for 28 days (as detected by blood smear analysis) following CHMI. | 28 days post each CHMI

SECONDARY OUTCOMES:
Antibody titers to Pf proteins by ELISA | Screening until week 52
  Assess the cellular and antibody responses induced by the PfSPZ Vaccine to determine whether any immune response(s) correlate with protection.
Antibody titers to Pf parasite stages by IFA | Screening until week 52
  Assess the cellular and antibody responses induced by the PfSPZ Vaccine to determine whether any immune response(s) correlate with protection.
Capacity to inhibit sporozoite invasion of hepatocytes in vitro by ISI assay | Screening until week 52
  Assess the cellular and antibody responses induced by the PfSPZ Vaccine to determine whether any immune response(s) correlate with protection.
Analysis of antibodies to any of the thousands of proteins in the Pf proteome using proteome array chips | Screening until week 52
  Assess the cellular and antibody responses induced by the PfSPZ Vaccine to determine whether any immune response(s) correlate with protection.
Multi-channel intracellular staining (ICS) analysis by flow cytometry against PfSPZ and synthetic peptides and recombinant proteins from defined Pf proteins | Screening until week 52
  Assess the cellular and antibody responses induced by the PfSPZ Vaccine to determine whether any immune response(s) correlate with protection.
Analysis of ELISpot responses in response to stimulation with PfSPZ and synthetic peptides and recombinant proteins from defined Pf proteins | Screening until week 52
  Assess the cellular and antibody responses induced by the PfSPZ Vaccine to determine whether any immune response(s) correlate with protection.
Analysis of T cell receptor studies | Screening until week 52
  Assess the cellular and antibody responses induced by the PfSPZ Vaccine to determine whether any immune response(s) correlate with protection.
B cell/plasmablast studies | Screening until week 52
  Assess the cellular and antibody responses induced by the PfSPZ Vaccine to determine whether any immune response(s) correlate with protection.
Human gene expression profiling focusing on immune response genes | Screening until week 52
  Assess the cellular and antibody responses induced by the PfSPZ Vaccine to determine whether any immune response(s) correlate with protection.
Luminex or Luminex type studies to assess multiple cytokines and other host molecules | Screening until week 52
  Assess the cellular and antibody responses induced by the PfSPZ Vaccine to determine whether any immune response(s) correlate with protection.

CONTACTS AND LOCATIONS:
Overall Officials: Judith Epstein, MD, Principal Investigator — Naval Medical Research Center
Locations (1):
- Walter Reed Army Institute of Research (WRAIR) Clinical Trials Center, Silver Spring, Maryland, United States

REFERENCES:
- [Result] Epstein JE, Paolino KM, Richie TL, Sedegah M, Singer A, Ruben AJ, Chakravarty S, Stafford A, Ruck RC, Eappen AG, Li T, Billingsley PF, Manoj A, Silva JC, Moser K, Nielsen R, Tosh D, Cicatelli S, Ganeshan H, Case J, Padilla D, Davidson S, Garver L, Saverino E, Murshedkar T, Gunasekera A, Twomey PS, Reyes S, Moon JE, James ER, Kc N, Li M, Abot E, Belmonte A, Hauns K, Belmonte M, Huang J, Vasquez C, Remich S, Carrington M, Abebe Y, Tillman A, Hickey B, Regules J, Villasante E, Sim BKL, Hoffman SL. Protection against Plasmodium falciparum malaria by PfSPZ Vaccine. JCI Insight. 2017 Jan 12;2(1):e89154. doi: 10.1172/jci.insight.89154. PMID 28097230